CLINICAL TRIAL: NCT00095277
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study of Darbepoetin Alfa Administered Once Every 4 Weeks in the Treatment of Subjects With Anemia of Cancer
Brief Title: Darbepoetin Alfa Administered Once Every 4 Weeks in the Treatment of Subjects With Anemia of Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20030204
Record Dates: First submitted 2004-11-02; First posted 2004-11-03 (Estimated); Last update posted 2009-03-13 (Estimated); Status verified 2009-03

CONDITIONS: Anemia
Keywords: non-myeloid malignancies; myeloma; Anemia of Cancer
MeSH Terms: conditions — Anemia; Neoplasms, Plasma Cell | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin Alfa

SUMMARY:
The purpose of this trial is to demonstrate benefit with respect to hematopoietic response in subjects with anemia of cancer randomized to Darbepoetin Alfa once every 4 weeks.

ELIGIBILITY:
Eligibility Criteria: - Subjects with non-myeloid malignancies - Subjects can not be on chemotherapy - Anemia of cancer - Eastern Cooperative Oncology Group (ECOG) status of 0 to 2 - Hemoglobin less than or equal to 11.0 g/dL - Adequate renal and liver function - Written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220
Dates: Start 2004-10

PRIMARY OUTCOMES:
To demonstrate benefit with respect to hematopoietic response in subjects with anemia of cancer randomized to darbepoetin alfa once every 4 weeks.

SECONDARY OUTCOMES:
Assess efficacy
Assess PROs
Assess relationship between PROs and hemoglobin concentration
Assess safety of dose and frequency

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Gordon D, Nichols G, Ben-Jacob A, Tomita D, Lillie T, Miller C. Treating anemia of cancer with every-4-week darbepoetin alfa: final efficacy and safety results from a phase II, randomized, double-blind, placebo-controlled study. Oncologist. 2008 Jun;13(6):715-24. doi: 10.1634/theoncologist.2007-0241. PMID 18586927
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_33_NESP_20030204.pdf
- See also: FDA-approved Drug Labeling — http://www.aranesp.com/